CLINICAL TRIAL: NCT03658317
Title: Renal Resisitive Index as an Indicator of the Progression of Diabetic Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, radwa awad abd elhafiz ibrahim, doctor ,assisstant lecturer,principle investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RI in diabetic nephropathy
Record Dates: First submitted 2018-09-01; First posted 2018-09-05 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases (Active Comparator): laboratory tests including (random blood glucose , serum urea and creatinine , lipogram , serum uric acid , HbA1c , urine analysis , 24 hours urinary proteins ) abdominal ultrasonography dupplex on the renal vessels
  Interventions: Diagnostic Test: renal arterial resistive index; Diagnostic Test: uric acid level; Diagnostic Test: serum urea and creatinine; Diagnostic Test: 24 hours urinary proteins; Diagnostic Test: lipogram; Diagnostic Test: HbA1c level; Diagnostic Test: urine analysis; Diagnostic Test: abdominal ultrasonography
- controls (Active Comparator): laboratory tests including (random blood glucose , serum urea and creatinine , lipogram , serum uric acid , HbA1c , urine analysis , 24 hours urinary proteins ) abdominal ultrasonography dupplex on the renal vessels
  Interventions: Diagnostic Test: renal arterial resistive index; Diagnostic Test: uric acid level; Diagnostic Test: serum urea and creatinine; Diagnostic Test: 24 hours urinary proteins; Diagnostic Test: lipogram; Diagnostic Test: HbA1c level; Diagnostic Test: urine analysis; Diagnostic Test: abdominal ultrasonography

INTERVENTIONS:
Diagnostic Test: renal arterial resistive index — done by dupplex on renal arteries
Diagnostic Test: uric acid level — serum sample for doing the test
Diagnostic Test: serum urea and creatinine — serum samples for doing the test
Diagnostic Test: 24 hours urinary proteins — urine collected over 24 hours for doing the test
Diagnostic Test: lipogram — serum sample for doing the test
  Other Names: lipid profile
Diagnostic Test: HbA1c level — serum sample for doing the test
Diagnostic Test: urine analysis — urine sample for doing the test
Diagnostic Test: abdominal ultrasonography — done by the ultrasonography device

SUMMARY:
diabetic nephropathy is one of the leading causes of end stage renal disease

DETAILED DESCRIPTION:
Diabetes mellitus is one of the systemic diseases affecting the kidneys. Diabetic nephropathy is a serious microvascular complication of diabetes mellitus. It is the most important cause of death in type I diabetic patients, of whom 30%-40% eventually develop end-stage renal failure and 40% of type II diabetics are at risk of developing diabetic nephropathy. So, diagnosis of diabetic nephropathy is paramount for the survivability of the diabetic patients not only because of the consequences of renal progression but also because of the strong association with the risk of developing cardiovascular disease Diabetic nephropathy (DN) is defined as persistent proteinuria greater than 500 mg/24 h, or albuminuria greater than 300 mg/24 h.

In the kidney, renal pathological changes leading to diabetic nephropathy are mainly secondary to atherosclerosis of the intra and extra renal arteries together with microangiopathy of the glomerular capillaries, afferent arterioles and efferent arteriole.

Doppler sonography may be a useful complementary test in the evaluation of DN, even in the early stages. Early stage of vascular involvement seems, in fact, to be characterized by functional alterations of endothelial control on vascular tone and wall interaction with circulating cells. Renal Doppler assessment of RI is a reliable, non-invasive evaluation of arterial function and is particularly useful for early diagnosis of vascular involvement.

Increasing evidence suggests that the intra-renal arterial RI, measured by Doppler ultrasound, a well-established technique for the investigation of renal morphology and hemodynamics, predicts the course of renal function in several conditions.

No standard, validated, cut-off to distinguish normal from high RI has been identified to date. RI values between 0.75 and 0.85 have been associated with renal functional impairment in patients with chronic kidney disease and stenosis of the renal artery, and they also predict allograft dysfunction in kidney transplant recipients Little information is available on the use of RI for the identification and prediction of DN in routine clinical practice. It is yet unclear whether RI predicts DN in low-risk patients; also, the correlation between increased intra-renal RI and altered renal hemodynamics remains unclear independent of albuminuria, as also the most appropriate cut-off value The renal arterial resistive index (RI) is a sonographic index to assess for renal arterial disease. It is measured as RI = (peak systolic velocity - end diastolic velocity ) / peak systolic velocity Measured at arcuate arteries (at the corticomedullary junction) or interlobar arteries (adjacent to medullary pyramids) intrarenal resistive index (RI) has been reported to be increased in hypertensive subjects with microalbuminuria and limited data is present for diabetic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients either type I or type II diabetes mellitus with or without any clinical evidence of diabetic nephropathy

Exclusion Criteria:

* Any disease affecting the cardiovascular system as vasculitis and hypertension Patients with ESRD due to diabetic nephropathy on regular dialysis Patients with nephrolithiasis Patients having any type of glomerulonephritis Patients with renal artery stenosis Renal transplantation recipients patients suffering from polycystic kidney disease or any other structural renal disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
renal resistive index | once(1day)
  calculated by the renal dupplex

SECONDARY OUTCOMES:
stage of diabetic nephropathy | once(1day)
  assessed by the proteinuria level

REFERENCES:
- [Background] Steinke JM, Mauer M; International Diabetic Nephropathy Study Group. Lessons learned from studies of the natural history of diabetic nephropathy in young type 1 diabetic patients. Pediatr Endocrinol Rev. 2008 Aug;5 Suppl 4:958-63. PMID 18806710
- [Background] Tublin ME, Bude RO, Platt JF. Review. The resistive index in renal Doppler sonography: where do we stand? AJR Am J Roentgenol. 2003 Apr;180(4):885-92. doi: 10.2214/ajr.180.4.1800885. No abstract available. PMID 12646425
- [Background] Youssef DM, Fawzy FM. Value of renal resistive index as an early marker of diabetic nephropathy in children with type-1 diabetes mellitus. Saudi J Kidney Dis Transpl. 2012 Sep;23(5):985-92. doi: 10.4103/1319-2442.100880. PMID 22982911
- [Result] Afsar B, Elsurer R. Increased renal resistive index in type 2 diabetes: Clinical relevance, mechanisms and future directions. Diabetes Metab Syndr. 2017 Oct-Dec;11(4):291-296. doi: 10.1016/j.dsx.2016.08.019. Epub 2016 Aug 30. PMID 27594114
- [Result] Gross JL, de Azevedo MJ, Silveiro SP, Canani LH, Caramori ML, Zelmanovitz T. Diabetic nephropathy: diagnosis, prevention, and treatment. Diabetes Care. 2005 Jan;28(1):164-76. doi: 10.2337/diacare.28.1.164. PMID 15616252
- [Result] Masulli M, Mancini M, Liuzzi R, Daniele S, Mainenti PP, Vergara E, Genovese S, Salvatore M, Vaccaro O. Measurement of the intrarenal arterial resistance index for the identification and prediction of diabetic nephropathy. Nutr Metab Cardiovasc Dis. 2009 Jun;19(5):358-64. doi: 10.1016/j.numecd.2008.07.003. Epub 2008 Sep 20. PMID 18805683
- [Result] Ozmen ND, Mousa U, Aydin Y, Deren T, Unlu EB. Association of the renal resistive index with microvascular complications in type 2 diabetic subjects. Exp Clin Endocrinol Diabetes. 2015 Feb;123(2):112-7. doi: 10.1055/s-0034-1390448. Epub 2014 Oct 24. PMID 25343266
- [Result] Shirin M, Sharif MM, Gurung A, Datta A. Resistive Index of Intrarenal Artery in Evaluation of Diabetic Nephropathy. Bangladesh Med Res Counc Bull. 2015 Dec;41(3):125-130. doi: 10.3329/bmrcb.v41i3.29888. PMID 29870167
- [Result] Said SM, Nasr SH. Silent diabetic nephropathy. Kidney Int. 2016 Jul;90(1):24-6. doi: 10.1016/j.kint.2016.02.042. PMID 27312444